CLINICAL TRIAL: NCT00922740
Title: An Open Label, Escalation Study to Assess Intra-Subject Dose Response to VA106483 in Elderly Male Subjects
Brief Title: VA106483 Dose Response Study in Elderly Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vantia Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 483-002
Record Dates: First submitted 2009-06-10; First posted 2009-06-17 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Nocturia
Keywords: Nocturia; Pharmacokinetics; Pharmacodynamics; Water-loading; Elderly; Males
MeSH Terms: conditions — Nocturia

ARMS (4):
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo
- VA106483 1 mg (Experimental)
  Interventions: Drug: VA106483
- VA106483 2 mg (Experimental)
  Interventions: Drug: VA106483
- VA106483 4 mg (Experimental)
  Interventions: Drug: VA106483

INTERVENTIONS:
Drug: VA106483 — Placebo on Day 1, 1 mg VA106483 on Day 3, 2 mg VA106483 on Day 5 and 4 mg VA106483 on Day 7
  Arms: VA106483 1 mg; VA106483 2 mg; VA106483 4 mg
Drug: Placebo — Placebo on Day 1, 1 mg VA106483 on Day 3, 2 mg VA106483 on Day 5 and 4 mg VA106483 on Day 7
  Arms: Sugar pill

SUMMARY:
The main purpose of the study is to evaluate the way VA106483 enters and leaves the blood and tissues over time and how the drug acts on and in the body at various dose levels compared to placebo in the same volunteer.

DETAILED DESCRIPTION:
VA106483 is intended to be used as a treatment for patients suffering from nocturia (defined as waking to urinate at least once per night between periods of sleep). Nocturia is a condition that often worsens as sufferers get older. This may be due to an over-active bladder muscle, the bladder being able to hold less urine at night-time or over production of urine in the bladder at night.

The only antidiuretic approved for the treatment (in some countries) of nocturia is the peptide drug, desmopressin. However, as it can cause hyponatraemia in a proportion of patients above the age of 65 years it is contra-indicated in the elderly. This side-effect has not been observed with VA106483, making it potentially suitable for treating the elderly. The purpose of this study is to confirm that duration of action of VA106483 can be effectively controlled by dose and therefore that satisfactory clinical outcome in the treatment of nocturia can be achieved by individual dose titration.

Subjects will be water-loaded, dosed with either VA106483 or placebo and then urine production will be monitored to assess any anti-diuretic effect.

ELIGIBILITY:
Inclusion Criteria:

* Male, Age: 65 years and above
* Using adequate contraception
* Medical history without clinically significant pathologies; no evidence of serious pathology or disease
* Physical examination parameters without signs of serious disease
* No clinically significant ECG and lab safety tests (sodium must be within normal range)
* Willing and able to participate and provides written informed consent

Exclusion Criteria:

* Cardiac insufficiency; signs or symptoms suggestive of heart failure or requiring treatment with diuretics
* Supine arterial blood pressure higher than 170/100 mmHg or less than 105/60 mm Hg
* Presence of poorly controlled endocrine disorders
* Renal insufficiency, active hepatic and/or biliary disease
* Hyponatraemia. Serum sodium level must be within normal limits
* Syndrome of inappropriate antidiuretic hormone (ADH) secretion
* Symptoms suggestive of psychogenic or habitual polydipsia or of diabetes insipidus
* Known hypersensitivity to the IP or any constituent of the IP
* Use of any non-prescription preparation within 72 hours prior to study entry, with the exception of defined pain killers
* A history of alcohol abuse or drug addiction within the last 2 years
* Positive screen for HIV, hepatitis B or C
* Currently taking any diuretics or any concomitant medication known to be a cytochrome 3A4 inhibitor
* Other protocol defined eligibility criteria may apply.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Urine volume and osmolality and plasma PK assessments | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Schutz, Principal Investigator — Quintiles Phase I Services, Overland Park, KS
Locations (1):
- Quintiles Phase I Services, Overland Park, Kansas, United States